CLINICAL TRIAL: NCT06419283
Title: Evaluation of the Safety and Efficacy of Stenting for Chronic Middle Cerebral Artery Occlusion With Limb Dysfunction: a Prospective Study
Brief Title: Prospective Study on Safety and Efficacy of Stenting for Chronic Middle Cerebral Artery Occlusion With Limb Dysfunction
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Huizhou Municipal Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LLBA201952A
Record Dates: First submitted 2024-05-07; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Chronic Middle Cerebral Artery Occlusion; Stenting Treatment; Modified Rankin Scale; National Institutes of Health Stroke Scale
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stenting group (Experimental): Middle Cerebral Artery Stent Implantation
  Interventions: Procedure: Middle Cerebral Artery Stent Implantation; Drug: standard treatment with aspirin.
- control group (Placebo Comparator): standard treatment with aspirin.
  Interventions: Drug: standard treatment with aspirin.

INTERVENTIONS:
Procedure: Middle Cerebral Artery Stent Implantation — Middle Cerebral Artery Stent Implantation
  Arms: stenting group
Drug: standard treatment with aspirin. — standard treatment with aspirin.

SUMMARY:
The goal of this clinical study is to evaluate the safety and efficacy of stenting for revascularization treatment of chronic middle cerebral artery (MCA) occlusion in patients with chronic MCA occlusion.

The main questions it aims to answer are:

1. Whether stenting treatment can improve blood flow restoration in chronic MCA occlusion.
2. If stenting can reduce the rates of reocclusion.
3. How stenting affects the recovery of neurological functions in these patients.

Researchers will compare the stenting group, which received stenting revascularization in addition to aspirin treatment, to the control group, which received only aspirin treatment to see if stenting treatment provides superior outcomes in terms of neurological function improvement and safety profile.

Participants will:

1. Undergo full cerebral angiography to identify the occlusion site.
2. All participants will be monitored for post-procedure complications and neurological function using the Modified Rankin Scale (mRS) and National Institutes of Health Stroke Scale (NIHSS) before and after treatment.
3. Participants will be followed up for three months post-treatment to assess the long-term efficacy and safety of the stenting procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age and gender: individuals aged 18 and above, regardless of gender.
* Diagnosis: chronic MCA occlusion confirmed by imaging studies (such as Magnetic Resonance Imaging (MRI) or Computed Tomography (CT)) for more than 3 months.
* Symptoms: neurological deficits caused by MCA occlusion, such as hemiplegia, speech disorders, etc.
* Treatment History: no stenting revascularization for MCA occlusion within the past three months.

Exclusion Criteria:

* Acute stroke: occurrence of an acute cerebrovascular event within the past three months.
* Other significant diseases: such as severe heart disease, liver or kidney dysfunction, cerebral hemorrhage, active bleeding, or coagulation disorders.
* Allergy to contrast agents.
* Severe mental illness or inability to comply with study requirements.
* Pregnant or breastfeeding women.
* Discovery of MCA occlusion without any symptoms.
* Participation in other clinical trials within the past six months.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
the Modified Rankin Scale (mRS) scores | 3 months
  The Modified Rankin Scale (mRS) scores serve as a critical outcome measure to assess the effectiveness of stenting treatment for patients with chronic middle cerebral artery (MCA) occlusion. The mRS is a standardized instrument that evaluates the degree of disability or dependence in daily activities following a stroke. It ranges from 0 (no symptoms) to 6 (death), with a higher mRS score indicates a greater level of disability or dependence.
the National Institutes of Health Stroke Scale (NIHSS) scores | 3 months
  The National Institutes of Health Stroke Scale (NIHSS) scores：By quantifying the degree of neurological deficits in stroke patients before and three months after surgery, the efficacy and safety of stent implantation can be assessed. The NIHSS score includes multiple items, with higher scores indicating more severe functional impairments, ranging from a total score of 0 (no stroke) to 42 (severe stroke).

CONTACTS AND LOCATIONS:
Locations (1):
- Huihong Huang, Huizhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT06419283/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT06419283/ICF_001.pdf